CLINICAL TRIAL: NCT01248403
Title: A Randomized, Double-blind, Multi-center Phase III Study Evaluating Paclitaxel With and Without RAD001 in Patients With Gastric Carcinoma Who Have Progressed After Therapy With a Fluoropyrimidine-containing Regimen
Brief Title: A Randomized, Double Blind Study Evaluating Paclitaxel With and Without RAD001 in Patients With Gastric Carcinoma After Prior Chemotherapy
Acronym: AIO-STO-0111
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Principal Investigator, Prof. Dr. S.E. Al-Batran, Principal Investigator, Krankenhaus Nordwest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRAD001RDE35T
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Advanced Gastric Cancer; Esophagogastric Junction Cancer
Keywords: RAD001; Paclitaxel; gastric cancer; advanced gastric or esophagogastric junction cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paclitaxel + placebo (Active Comparator): Paclitaxel 80 mg/m2 on day 1, day 8 and day 15 of every 28-day cycle.
  + Placebo (2 tablets / day) d1-d28
  Interventions: Drug: Paclitaxel
- paclitaxel + RAD001 (Experimental): Paclitaxel 80 mg/m2 on day 1, day 8 and day 15 of every 28-day cycle.
  + RAD001 10mg (2 x5 mg tablets / day) d1-d28
  Interventions: Drug: Paclitaxel; Drug: RAD001

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 80 mg/m2 on day 1, day 8 and day 15 of every 28-day cycle.
Drug: RAD001 — RAD001 10mg (2 x5 mg tablets / day) d1-d28
  Other Names: Everolimus; Certican
  Arms: paclitaxel + RAD001

SUMMARY:
Adult patients with gastric carcinoma which has progressed after initial treatment with a fluoropyrimidines-containing regimen will be treated with paclitaxel plus RAD001 or plus placebo. The hypothesis is that patients with RAD001 have significantly prolonged overall survival compared to patients who are treated with paclitaxel alone.

DETAILED DESCRIPTION:
This is a randomized, double-blind, phase III two-arm multi-center study aiming at estimating the relative efficacy of the combination of RAD001 and paclitaxel versus that of paclitaxel alone as second-, third- or fourth-line treatment in terms of hazard ratio of overall survival in patients with gastric cancer who have relapsed after one treatment regimen containing a fluoropyrimidine (e.g., 5-FU, S-1, capecitabine and other 5-FU prodrugs or derivatives). Patients will be randomized in a 1:1 ratio for a total of 240 patients per treatment arm. Randomization will be stratified according to performance status (0-1 versus 2), prior taxan use (yes vs. no) and treatment line (2nd versus 3rd/4th line).

Study treatment will be continued until progression or intolerable toxicity. Patients will be seen at baseline/screening, and weekly for paclitaxel administration and safety assessment until disease progression or discontinuation of trial therapy for other reasons. Radiological tumor assessment will be performed every second cycle (every 8 weeks) or earlier if clinically indicated. Post-study follow-up will be completed every 8 weeks for survival.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years old
* Histologically or cytologically confirmed and documented gastric adenocarcinoma. Adenocarcinomata of the gastro-esophageal junction will be allowed, if they have advanced disease (inoperable, recurrent or metastatic disease).
* Documented progressive disease during/after one, two or three prior treatments containing 5FU and/or its precursors or derivatives in the palliative setting
* At least one measurable or evaluable lesion by RECIST as determined by Computed Tomography (CT) Scan or Magnetic Resonance Imaging (MRI)
* ECOG performance status of 0, 1 or 2
* The following laboratory parameters:

  * Absolute neutrophil count ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Serum creatinine ≤ 2 x Upper Limit of Normal (ULN)
  * Adequate liver function:
  * Total serum calcium (corrected for serum albumin) or ionized calcium ≥ LLN
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of the first administration of study treatments and must be willing to use adequate methods of contraception during the study and for 3 months after last study drug administration.
* Written informed consent

Exclusion Criteria:

* Current treatment with any anti cancer therapy or treatment with anti cancer therapy ≤ 2 weeks prior to study treatment start unless rapidly progressing disease is measured
* Known hypersensitivity to RAD001 (everolimus) or to its excipients, or to other rapamycins (e.g. sirolimus, temsirolimus)
* Known prior history of hypersensitivity to paclitaxel.
* Paclitaxel refractory disease, which is defined as a disease progression under or within 12 weeks of last taxan treatment
* Chronic treatment with steroids (except for oral, topical or local injection) or another immunosuppressive agent
* Major surgery ≤ 2 weeks prior to starting study treatment or patients who have not recovered from such therapy
* Lack of resolution of all acute toxic effects (excluding alopecia) of prior chemotherapy, prior radiotherapy, or surgical procedure to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade <= 1. Note: Neuropathy due to prior chemotherapy is allowed.
* Unstable CNS disease

  * Requiring increasing doses of steroids to maintain stable neurological status
  * Deteriorating / changing neurological status
* Known history of HIV seropositivity (HIV testing is not mandatory) or Hepatitis B or C.
* Active, bleeding diathesis or on oral anti-vitamin K medication (except low dose warfarin, as long as the INR is <= 2.0)
* Any other severe and/or uncontrolled medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
overall survival | 6 months follow-up

SECONDARY OUTCOMES:
best overall response | staging every 8 weeks
progression-free survival | staging every 8 weeks
number of participants with adverse events as a measure of safety and tolerability | every week until end of treatment
disease control rate | every 8 weeks
  responders + stable disease ≥12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, MD, Principal Investigator — Institute of Clinical Cancer Research (IKF), UCT - University Cancer Center, Frankfurt, Germany
Locations (1):
- Krankenhaus Nordwest, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Lorenzen S, Knorrenschild JR, Pauligk C, Hegewisch-Becker S, Seraphin J, Thuss-Patience P, Kopp HG, Dechow T, Vogel A, Luley KB, Pink D, Stahl M, Kullmann F, Hebart H, Siveke J, Egger M, Homann N, Probst S, Goetze TO, Al-Batran SE. Phase III randomized, double-blind study of paclitaxel with and without everolimus in patients with advanced gastric or esophagogastric junction carcinoma who have progressed after therapy with a fluoropyrimidine/platinum-containing regimen (RADPAC). Int J Cancer. 2020 Nov 1;147(9):2493-2502. doi: 10.1002/ijc.33025. Epub 2020 May 7. PMID 32339253